CLINICAL TRIAL: NCT03892655
Title: A Multicenter, Prospective, Real World, National Study to Assess the Efficacy and Safety of Adjuvant Biosimilar Tratuzumab (Zedora) Treatment in Patients With Localized Her2 Positive Breast Cancer
Brief Title: Real World Study of Biosimilar Trastuzumab in Her2 Positive Breast Cancer
Acronym: LB1802
Status: Active, not recruiting | Type: Observational
Sponsor: Libbs Farmacêutica LTDA (Industry)
Responsible Party: Sponsor
Other Study IDs: LB1802
Record Dates: First submitted 2019-02-12; First posted 2019-03-27 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: breast carcinoma; receptors 2 (HER2); biosimilar; trastuzumab; Zedora
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Zedora registration was based on studies of women with metastatic breast cancer, but its approval includes adjuvant treatment. Thus, prospective data of drug use in localized disease are lacking, as well as are real-world safety and efficacy data, taking into consideration comorbidities and compliance difficulties.

This will be an observational study of patients receiving adjuvant Zedora at several Brazilian institutions for the purpose of describing its efficacy and safety.

DETAILED DESCRIPTION:
An observational, multicenter, prospective, real-world study at Brazilian institutions.

Adult patients with early HER2+ breast cancer receiving adjuvant biosimilar trastuzumab (Zedora) at the participating sites after the start of the study and meeting the eligibility criteria will be invited to participate. Demographics, comorbidities, disease history, extent of exposure to biosimilar trastuzumab (Zedora), adverse events and LVEF values will be collected.

Data collection will be performed using a case report form (CRF) specifically designed for the study.

Study Treatment:

Biosimilar trastuzumab (Zedora) must be prescribed at the dosage described in the product label.

Treatment duration will be 12 months for patients starting upfront with biosimilar trastuzumab (Zedora). Patients switching at any time to biosimilar trastuzumab (Zedora) after a period of adjuvant or neoadjuvant Herceptin® use will also be included in the overall analysis and subsequently assessed in a subgroup analysis.

Sample Size:

Number of patients = 170 Given the inexistence of a specific hypothesis to be tested, the statistical analysis will be basically descriptive.

Sample size is based on the two-sided 95% confidence interval (95% CI) for the invasive disease relapse-free survival rate.

The table below shows the 95% CIs for different rates in a sample of 170 patients, with an interval size ranging between 9% and 15%.

Based on literature, a 3-year relapse-free survival between 88 and 96% is expected. According to the table above, a sample of 170 patients allows assessing this endpoint with +/- 6.0% accuracy.

Study duration:

The estimated time for patient enrollment in the study is one year and may be extended in case the sample size is not reached in this period. Biosimilar trastuzumab (Zedora) must be prescribed according to the product label and treatment duration will be up to one year. The patient will be maintained in the study for 5 years (from start of treatment), unless there is tumor recurrence (local or distant).

ELIGIBILITY:
Inclusion Criteria:

* female patients aged 18 years and over
* diagnosis of early stage I to III breast cancer confirmed by histopathology test according to local guidelines.
* human epidermal growth factor receptor 2 (HER2)-positive tumor by immunohistochemistry or FISH (Fluorescence In Situ Hybridization), as per the 2018 ASCO assessment guideline [J Clin Oncol 36:2105, 2018].
* use of at least one dose of biosimilar trastuzumab (Zedora) as adjuvant therapy, regardless of previous neoadjuvant trastuzumab or Zedora use or the type of chemotherapy combined with the antibody.
* Signing of the informed consent form (ICF).

Exclusion Criteria:

* use of biosimilar trastuzumab (Zedora) differently from the provisions in the label.
* patients enrolled in and followed up by Programa Vida Plena [Full Life Program].

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult female patients with diagnosis of early stage I to III HER2+ breast cancer confirmed by histopathology test, immunohistochemistry test and FISH, where required, according to local guidelines, and who have started biosimilar trastuzumab (Zedora) as neoadjuvant or adjuvant therapy according to the product label will be eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Efficacy endpoints: Invasive disease relapse-free survival rate | 18 months
  Invasive disease relapse-free survival rate
Efficacy endpoints: Invasive disease relapse-free survival rate | 24 months
  Invasive disease relapse-free survival rate
Efficacy endpoints: Invasive disease relapse-free survival rate | 30 months
  Invasive disease relapse-free survival rate
Efficacy endpoints: Invasive disease relapse-free survival rate | 36 months
  Invasive disease relapse-free survival rate
Efficacy endpoints: Invasive disease relapse-free survival after curative-intent surgery | 5 years
  Invasive disease relapse-free survival after curative-intent surgery
Efficacy endpoints: Overall survival after curative intent surgery | 5 years
  Overall survival after curative intent surgery
Safety endpoints: Incidence of Related Adverse Events | 5 years
  Incidence of Related Adverse Events
Safety endpoints: Total cycles per patient | 5 years
  Total cycles per patient
Safety endpoints: Incidence of dose interruption | 5 years
  Incidence of dose interruption

CONTACTS AND LOCATIONS:
Locations (22):
- Brazil (22):
  - William Hiromi Fuzita, Manaus, Amazonas
  - Márcia Cristina Colares Régis de Araújo, Fortaleza, Ceará
  - Raphael Luzorio Fernandes, Cachoeiro de Itapemirim, Espírito Santo
  - Sabina Bandeira Aleixo, Cachoeiro de Itapemirim, Espírito Santo
  - Daniel Fontes Santos de Teive e Argolo, Salvador, Estado de Bahia
  - Ruffo de Freitas Junior, Goiânia, Goiás
  - Cristina de Deus Anjos Tavares Sampaio, Campo Grande, Mato Grosso
  - Luis Eduardo Rosa Zucca, Três Lagoas, Mato Grosso do Sul
  - Micheline Campos Rezende, Muriaé, Minas Gerais
  - Karina Costa Maia Vianna, Curitiba, Paraná
  - Sérgio Lunardon Padilha, Curitiba, Paraná
  - Sâmio Pimentel Ferreira, Belém, Pará
  - Cláudio Rocha, Teresina, Piauí
  - Andrea Juliana Pereira de Santana Gomes, Natal, Rio Grande do Norte
  - Tomas Reinert, Caxias do Sul, Rio Grande do Sul
  - Rafaela Kirchner Piccoli, Ijuí, Rio Grande do Sul
  - Mateus Bongers Alessandretti, Porto Alegre, Rio Grande do Sul
  - Charles Alain Cordova Pinto, Lages, Santa Catarina
  - Daniel Grabarz, Mogi das Cruzes, São Paulo
  - Monique Celeste Tavares, São Paulo, São Paulo
  - Kaique Almeida, São Paulo, São Paulo
  - Mariana Scaranti, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gagliato D, Reinert T, Rocha C, Tavares M, Pimentel S, Fuzita W, Araujo M, Matias D, Aleixo S, Franca B, Magaton E, Brito N, Cardoso AC, Castilho V. Real-World Study of Adjuvant Biosimilar Trastuzumab-dkst for HER2-Positive Breast Cancer Treatment in a Brazilian Population. Oncol Ther. 2024 Sep;12(3):437-449. doi: 10.1007/s40487-024-00284-5. Epub 2024 Jun 5. PMID 38836997